CLINICAL TRIAL: NCT05121883
Title: An Observational Trial of Edaravone Dexborneol Combining With Mechanical Thrombectomy in the Treatment of Acute Ischemic Stroke
Brief Title: Edaravone Dexborneol Combining With Mechanical Thrombectomy in the Treatment of Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: EDMETS
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Edaravone dexborneol group: Patients with edaravone dexborneol initiating within 48 hours of stoke onset at 37.5 mg/dose, once every 12 hours, and continuing for more than 7 days will be classified into this group.
  Interventions: Drug: Edaravone Dexborneol
- Standard medication group: Patients who do not recieve edaravone dexborneol will be classified into this group.

INTERVENTIONS:
Drug: Edaravone Dexborneol — Edaravone dexborneol (Jiangsu Simcere Pharmaceutical, Co, Ltd) will be initiated within 48 hours of stoke onset at 37.5 mg/dose, once every 12 hours, and continuing for more than 7 days (maximum: 14 days)
  Groups: Edaravone dexborneol group

SUMMARY:
Edaravone dexborneol, comprised of 2 active ingredients, edaravone and (+)-borneol, has been developed as a novel neuroprotective agent with synergistic effects of antioxidant and anti-inflammatory in animal models. The TASTE trial (Treatment of Acute Ischemic Stroke with Edaravone Dexborneol) administered edaravone dexborneol or edaravone alone to stroke patients within 48 hours after stroke onset, finding that 90-d functional outcome was better in edaravone dexborneol group. However, the TASTE trial excluded patients undergoing reperfusion therapy (i.e., intravenous thrombolysis and mechanical thrombectomy). Therefore, the investigators aim to evaluate the efficacy of edaravone dexborneol in addition to mechanical thrombectomy in the treatment of acute ischemic stoke.

DETAILED DESCRIPTION:
This is a prospective, non-randomized clinical trial in multiple stroke centres of China. The total sample size will be 200. Patients with anterior-circulation large artery occlusion obtaining successful recanalization after mechanical thrombectomy (MT) will be assigned into edaravone dexborneol or standard medication treatment group based on whether or not receiving edaravone dexborneol. Only patients with edaravone dexborneol initiating within 48 hours of stoke onset at 37.5 mg/dose, once every 12 hours, and continuing for more than 7 days could be enrolled as edaravone dexborneol group. Patients in standard medication treatment group must not receive edaravone dexborneol. Other neuroprotective agents are not limited to use.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with anterior circulation acute ischemic stroke
* Patients aged between 18-80 years.
* CTA or DSA verified arterial occlusion of ICA, M1 or M2.
* NIHSS on admission 4 - 26
* Baseline CTP verified infarct core < 70 ml, penumbra > 10 ml, hypoperfusion/core > 1.8
* Undergoing mechanical thrombectomy within 24 hours of stroke onset. For wake-up stroke, the onset time is determined as the midpoint of last-seen-well and discovered time

Exclusion Criteria:

* Patients without recanalization (TICI 0,1, 2a)
* Pre-existing neurological disability (a score greater than 2 on the mRS)
* Contraindication of edaravone dexborneol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18-80 years with anterior circulation stroke obtaining successful recanalization after mechanical thrombectomy within 24 hours of onset will be included. CTP prior to mechanical thrombectomy must be performed to verify infarct core < 70 ml, penumbra > 10 ml, hypoperfusion/core > 1.8. Patients without recanalization after mechanical thrombectomy or have a pre-mRS greater than 2 will be excluded.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of functional independence at 90 days | 90 days
  Functional independence will be assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Growth in infarct volume (mL) | from 24 hours to 7 days
  24 hour infarct volume (mL) - 7 day infarct volume (mL)
Salvaged ischemic tissue index (%) | from baseline to 7 days
  100%*(baseline hypoperfusion (mL) - 7 day infarction lesion (mL))/ baseline hypoperfusion (mL)
Frequency of parenchymal hemorrhage (PH) (%) | 24 hours
  The presence of PH is defined according the standard from ECASS-2 study thrombectomy
Change on the National Institute of Health stroke scale (NIHSS) score from baseline to 1 day | from baseline to 1 day
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Change on the National Institute of Health stroke scale (NIHSS) score from 1 day to 7 day | from 1 day to 7 days
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Excellent recovery assessed by the ratio of modefied Rankin Scale (mRS) score of 0-1 | 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Recovery assessed by modefied Rankin Scale (mRS) score | 90 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, MD, Study Chair — the 2nd affiliated hospital of Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided